CLINICAL TRIAL: NCT07342816
Title: Exploring the Impact of Mindfulness on Athletic Performance and Functional Movement in Collegiate Athletes
Brief Title: Impact of Mindfulness on Athletic Performance and Functional Movement in Collegiate Athletes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Macau (Other)
Responsible Party: Principal Investigator, Siman Lei, Assistant Professor, University of Macau
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HE-1286-2025
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Athletic Performance; Mental Health
Keywords: Mindfulness; Athletic Performance; Collegiate Athletes; Basketball; Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness Intervention (MAIC) Group (Experimental): Participants assigned to this group receive an 8-week "Mindfulness-Acceptance-Insight-Commitment" (MAIC) program. The intervention is delivered in a "micro-dosing" format, consisting of 15-20 minute sessions conducted three times per week (Monday, Wednesday, Saturday) immediately before or after regular basketball training. The curriculum focuses on developing non-judgmental awareness, acceptance of internal states, and commitment to value-driven behavior to enhance psychological flexibility and performance.
  Interventions: Behavioral: Mindfulness-Acceptance-Insight-Commitment (MAIC) Program
- Psychological Skills Training (PST) Group (Active Comparator): Participants assigned to this group receive an 8-week Psychological Skills Training (PST) program serving as an active control. To ensure structural equivalence with the experimental arm, sessions are also 15-20 minutes long and conducted three times per week. The training covers traditional sports psychology techniques, including goal setting, imagery, arousal regulation, and positive self-talk.
  Interventions: Behavioral: Psychological Skills Training (PST) Program
- Control Group (No Intervention): Participants in this group receive no additional psychological intervention during the 8-week study period. They simply maintain their standard university basketball team training routine. After the completion of all study assessments, they are offered the opportunity to receive the mindfulness training program.

INTERVENTIONS:
Behavioral: Mindfulness-Acceptance-Insight-Commitment (MAIC) Program — Participants undergo an 8-week mindfulness training program based on the MAIC model developed by Si, Zhang, & Su (2019) . The program is adapted from the Mindfulness-Acceptance-Commitment (MAC) approach, incorporating an "Insight" component tailored for Asian culture . The intervention aims to reduce experiential avoidance and enhance psychological flexibility . It is delivered in a "micro-dosing" format consisting of three 15-20 minute sessions per week, integrated directly into regular basketball training schedules . Key components include mindfulness breathing, body scanning, values clarification, cognitive defusion, and acceptance strategies.
  Other Names: MAIC; Mindfulness Training
  Arms: Mindfulness Intervention (MAIC) Group
Behavioral: Psychological Skills Training (PST) Program — Participants undergo an 8-week systematic psychological skills training program serving as an active control. To ensure structural equivalence with the experimental arm, the dosage is matched at three sessions per week, each lasting 15-20 minutes. The curriculum covers traditional sports psychology techniques for self-regulation, including arousal regulation, goal setting, imagery (visualization), attentional control, cognitive restructuring (positive self-talk), and pre-performance routines.
  Other Names: PST; Mental Skills Training
  Arms: Psychological Skills Training (PST) Group

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of a mindfulness training program on sports performance and mental health in university basketball players. The main questions it aims to answer are:

1. Does the mindfulness program improve basketball skills, body movement control, and psychological health?
2. Does the program's effectiveness differ between male and female athletes?
3. Is there an association between athletes' current psychological states and their athletic performance before training?

Researchers will compare a mindfulness group to a psychological skills training group and a standard control group to see if the mindfulness program leads to significantly greater improvements in performance and well-being.

Participants will:

1. Complete surveys about their mental health and stress.
2. Perform physical fitness tests, such as jumping, running, and strength exercises.
3. Perform basketball skill tests, including shooting, dribbling, and passing.
4. Play in standardized 5-on-5 basketball games that are video-recorded for analysis .
5. Attend 15-to-20-minute training sessions 3 times a week for 8 weeks (if assigned to a training group) .

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be active university basketball athletes enrolled at the University of Macau, City University of Macau, or Macau University of Science and Technology .
2. Participants must be 18 years of age or older.
3. Participants must not have a current musculoskeletal injury or chronic condition that prevents participation in high-intensity physical assessments
4. Participants must not have significant prior experience with formal mindfulness or meditation practice.
5. Participants must not have received prior systematic Psychological Skills Training (PST) courses.
6. Participants must be able to commit to the 8-week intervention and assessment schedule.

Exclusion Criteria:

1. Individuals who do not meet the specific inclusion criteria (e.g., not a current university basketball athlete at the specified universities, or under 18 years old).
2. Presence of a musculoskeletal injury or chronic condition that prevents safe participation in physical assessments.
3. Significant prior experience with formal mindfulness or meditation practice, defined as having attended a course lasting one week or more.
4. Prior participation in systematic Psychological Skills Training (PST).
5. Inability to commit to the full 8-week intervention timeline.
6. Refusal to provide informed consent or declines to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Stationary Free-throw Accuracy | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  To evaluate the basic shooting accuracy without the influence of defensive pressure and fatigue, this study will adopt a standardized static free throw test. According to the process of Pojskic, Sisic, Separovic, & Sekulic (2018), after completing the designated warm-up procedure, participants will take three sets of free throws on the standard free-throw line, with 10 consecutive attempts in each set, and a complete 3-minute break between each set. During the test, two researchers will be responsible for picking up the backboard under the basket and quickly passing the ball back to the participants to maintain a stable test rhythm. The study will record and calculate the average shooting percentage of the participants in all three groups (a total of 30 shots), which will be used as a reference indicator to evaluate their basic free throw skills.
1-Minute Shooting Test | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  To quantify the shooting efficiency and stability of athletes under combined movement, this study will adopt a one-minute shooting test, and the specific process will refer to the research of Kumari, Singh, & Varghese (2023). Before the test, researchers will set shooting points at five angles of 0°, 45°, 90°, 135° and 180° at a distance of 4.54 meters from the center of the basket. After the test begins, a one-minute timer is set. Participants need to move their shots in a loop between five points. After each shot, regardless of whether it is successful or not, the participants must rush for the rebound by themselves and then dribble to the next position to shoot again. This test adopts a special scoring system: 2 points are awarded for each successful shot. A shot that misses but the ball touches the rim earns one point. The final score is the total score obtained by the participants within one minute.
Stationary 2-Point Shooting Accuracy | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  To evaluate the basic shooting accuracy at mid-range and without fatigue, this study will adopt a standardized static two-point shot test. According to the protocol of Pojskic, Sisic, Separovic, & Sekulic (2018), after standardized warm-up, participants will undergo three sets of shooting tests, with a complete 3-minute rest between each set. In each set of tests, participants need to take two jump shots from five different positions 5 meters away from the center point of the basket. That is, each group takes a total of 10 shots. The test will be conducted without any time limit, and two researchers will be responsible for picking up the backboard and passing the ball under the basket to ensure a smooth process. Ultimately, the study will record and calculate the average shooting percentage of the participants across all three groups (a total of 30 shots) as an indicator of their static two-point shooting ability.
Stationary 3-Point Shooting Accuracy | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  To evaluate the basic shooting accuracy at a long distance and without fatigue, this study will adopt a standardized static three-point shot test. To ensure methodological consistency, the process of this test is exactly the same as that of the static two-point shot test, with only the shooting distance changed to outside the standard three-point line (Pojskic, Sisic, Separovic, & Sekulic, 2018). Participants also need to complete three sets of tests. In each set, they take two shots from five different positions outside the three-point line (a total of 10 shots), with a three-minute break between sets. The test was also conducted without time limit, with two researchers assisting in passing the ball. Ultimately, the study will record and calculate the average shooting percentage of the participants across all three groups (a total of 30 shots) as an indicator of their static three-point shooting ability.
"I" Dribble Test | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  The site layout includes five marker cones: Cone 1 is 8 meters away from the starting line, Cone 2 to Cone 5 are placed every 3 meters in sequence, with the farthest distance being 20 meters. The test uses the Witty SEM, Microgate system for precise timing. The test process is as follows: The participant holds the ball and stands behind the starting line. Upon hearing the signal, they first dribble and sprint to Cone 1 and then return to the starting line. They then continue dribbling around Cone 1 to Cone 5, and finally dribble and sprint 20 meters in a straight line from Cone 5 back to the starting line. The timing ends. If the ball is lost during the process (the ball rolls more than two steps away from the body), this test is invalid. Each participant should complete two valid tests with at least a five-minute break in between. The shortest time (in seconds) will be taken as the final score.
Control Dribble Test | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  To assess the ball control ability of athletes on complex routes, this study will adopt the controlled dribbling test. According to the setup of Kumari, Singh, & Varghese (2023), researchers will use five marker cones to arrange a specific dribbling route within a 5.8-meter x 3.6-meter area. At the beginning of the test, participants need to dribble the ball with their non-dominant hand and go around all the marker cones as quickly as possible along the preset complex route. The entire process will use a timer to record the time (in seconds) required to complete the entire course. Each participant will take three tests, and the one with the shortest time taken will be the final score.
CODAT with Ball | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  This study will adopt the ball-holding Direction Change Acceleration Test (CODAT) (Puente et al., 2017). Before the test, researchers will use marker cones to lay out a standardized route. The test will use the electronic timing gate system (Witty SEM, Microgate, Bolzano, Italy) for precise timing. Participants hold the ball and stand behind the starting line. Upon hearing the signal, they complete the designated route at the fastest speed, including forward dash, sudden stop, 45-degree and 90-degree turn dribbling, etc. Throughout the entire process, participants must always maintain control of the ball. If a goal is conceded or the test is not completed along the prescribed route during the process, the test will be invalid. Each participant will take two tests, with at least a three-minute complete break in between. The shortest recorded time (in seconds) will be taken as the final score.
Linear Sprints with Dribbling | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  To measure the maximum speed of an athlete when dribbling and advancing with full force without the interference of changing direction, this study will adopt a 20-meter straight-line sprint test with the ball. This test also uses an electronic timing gate system. A pair of photoelectric sensors are set at the starting point and the 20-meter finish line respectively to ensure the accuracy of the data (Scanlan et al., 2019). Participants start from a position 30 centimeters behind the starting line with the ball in hand. Upon hearing the signal, they dribble forward with all their might and sprint forward. The study will record the time (in seconds) required for participants to complete the entire 20-meter course. Each participant will take two valid tests, with at least a three-minute complete break in between. The shortest recorded time will be taken as the final score.
Wall Passing Test | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  Participants perform chest passes against a wall with 6 target squares (3 high, 3 low) from a 2.5m distance for 30 seconds, using slide steps to move between targets. Scoring: 2 points for hitting the target, 1 point for hitting the wall between targets.
In-Game Performance Statistics | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  Performance in a standardized 5-on-5 full-court game is recorded by two independent observers. Statistics (points, rebounds, assists, steals, blocks, fouls, turnovers, etc.) are converted into a Performance Index Rating (PIR) using the FIBA formula.
Change in Functional Movement Control | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  Assessed using the Functional Movement Screen (FMS™). This tool evaluates seven fundamental movement patterns: Deep Squat, Hurdle Step, Inline Lunge, Shoulder Mobility, Active Straight-Leg Raise, Trunk Stability Push-up, and Rotary Stability. Each pattern is scored from 0 to 3 based on execution quality and pain presence, with a maximum total score of 21.
Athlete Psychological Strain Questionnaire (APSQ) | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  The APSQ consists of 10 items, aiming to quickly assess the degree of psychological tension and distress of athletes in sports-related situations (such as "In the past four weeks, I couldn't stop worrying about injuries or performance"). Participants are required to rate the frequency of each item based on their feelings over the past four weeks using a five-point Likert scale (1= never, 5= always). The scoring method is to directly add up the scores of all items, with the total score ranging from 10 to 50 points. According to the official guidelines of SMHAT-1, if the total score is equal to or higher than 17 points, it indicates that the athlete may have a relatively high risk of psychological distress and requires further attention or assessment. The Chinese version of this tool has been verified for reliability and validity among Chinese elite athletes (HKSI, 2021).
Beck Anxiety Inventory, BAI | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  The BAI scale consists of 21 items and requires participants to rate the severity of each anxiety symptom (such as "accelerated heartbeat", "fear", "tension", etc.) based on their feelings over the past week. The scale is scored using the Likert four-point scale (0= none, 1= mild, 2= moderate, 3= severe), and the total score is the sum of the scores of all items, ranging from 0 to 63 points. According to the standard interpretation, a score of 0 to 7 indicates extremely mild anxiety, 8 to 15 indicates mild anxiety, 16 to 25 indicates moderate anxiety, and 26 to 63 indicates severe anxiety. BAI is a widely used anxiety assessment tool in clinical practice and research. Its Chinese version has been proven to have excellent reliability and validity. In the study conducted by Zheng Yuyu et al. (2002) on a Taiwanese community sample, its internal consistency reliability (Cronbach's α) was as high as 0.94.
Sport Anxiety Scale-2, SAS-2 | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  SAS-2 consists of 15 items and is scored using the Likert Four-point Scale (1= not at all, 4= very serious), with a total score ranging from 15 to 60 points. This scale can assess competitive Trait Anxiety from three core dimensions: (a) Somatic Trait Anxiety, which includes five items, is used to measure the physiological tension responses (such as accelerated heart rate and muscle tightness) that athletes usually feel during competitions; (b) Worry, which consists of five items, is used to measure the degree of athletes' concern about their own poor performance and negative evaluations from others; And (c) Concentration Disruption, which consists of five items, is used to measure the tendency of athletes to have difficulty concentrating during competitions. The Chinese version of SARS-2 also demonstrated excellent psychometric characteristics among the Chinese athlete community, with an internal consistency reliability (Cronbach's α) of.89 (Huang Chongru, 2009).
Beck Depression Inventory-II, BDI-II | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  This scale consists of 21 items, each corresponding to a specific category of depressive symptoms (such as "sadness", "loss of interest", "fatigue", etc.). Participants are required to select the most appropriate sentence from each group of four statements describing different degrees of severity based on their feelings over the past two weeks. The scale is scored on a four-point scale (0 to 3 points), with the total score being the sum of all item scores, ranging from 0 to 63 points. According to the standard interpretation, a score of 0 to 13 indicates no or very mild depression, 14 to 19 indicates mild depression, 20 to 28 indicates moderate depression, and 29 to 63 indicates severe depression. The Chinese version of BDI-II has been widely used and has proved to have excellent reliability and validity. In the study conducted by The Chinese University of Hong Kong (2005), the internal consistency reliability (Cronbach's α) of the Chinese version was as high as 0.92.
Perceived Stress Scale, PSS-10 | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  This study adopted its simplified version (PSS-10) consisting of 10 items, asking participants to assess the frequency of specific feelings or thoughts occurring in the past month. The scale is scored using the Likert five-point scale (0= never, 4= very frequent). Among them, the four items with positive expressions (#4, 5, 7, 8) need to be processed in reverse when scoring. The total score is obtained by adding up the scores of all items, ranging from 0 to 40 points. The higher the score, the higher the perceived stress level of the individual. Its reliability and validity were good in the Chinese sample. In the study in Taiwan region, the internal consistency reliability (Cronbach's α) of the Chinese version of PSS-10 was.85 (Chu, 2010).
Recovery-Stress Questionnaire for Athletes, RESTQ-Sport | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  This study adopts a version consisting of 76 items, corresponding to 19 different sub-dimensions (with 4 items in each sub-dimension). These sub-dimensions can be classified into two major categories: general stress dimensions (such as "general stress", "emotional exhaustion", "injury"), general recovery dimensions (such as "success", "physical recovery", "sleep quality"), specific stress dimensions (such as "training stress", "competition anxiety"), and specific recovery dimensions (such as "personal responsibility", "self-efficacy"). Participants are required to assess the frequency of their feelings over the past three days based on the Likert seven-point scale (0= never, 6= always). The scoring method is to calculate the average score of the 19 sub-dimensions respectively, thereby providing a detailed profile of the athlete's current stress-recovery status.
Athlete Burnout Questionnaire, ABQ | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  The ABQ consists of 15 items and is scored using the Likert five-point Scale (1= almost never, 5= almost always). These three dimensions are evaluated respectively: (a) Emotional/Physical Exhaustion, which consists of five items, is used to measure the fatigue and energy depletion that athletes feel due to training and competition; (b) Reduced Sense of Accomplishment, which consists of five items, is used to measure the tendency of athletes to negatively evaluate their athletic ability and achievements; And (c) Sport Devaluation, which consists of five items, is used to measure athletes' negative and cynical attitudes towards the meaning and value of the sports they are engaged in. When scoring, the average score of each of the three sub-dimensions is calculated separately. The higher the score, the more severe the degree of burnout in that dimension. The internal consistency reliability (α) of each subscale of the original scale ranged from.89 to.93.

SECONDARY OUTCOMES:
Five-Facet Mindfulness Questionnaire (FFMQ) | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  This scale consists of 39 items, corresponding to five sub-dimensions respectively: (a) Observing; (b) Describing; (c) Acting with Awareness; (d) Non-judging of Inner Experience; And (e) Non-reactivity to Inner Experience. Participants are required to rate the description of each item based on the Likert five-point scale (1= completely inconsistent, 5= completely consistent). The total score ranges from 39 to 195 points. The higher the total score and the scores of each sub-dimension, the higher the level of mindfulness traits of the individual in the corresponding aspect. This scale has been translated and subjected to rigorous psychometric tests in Chinese samples. The research by Deng Yuangui et al. (2012) shows that the Chinese version of FFMQ has good internal consistency reliability. The Cronbach's α coefficient of its total scale is.88, and the α coefficients of each subscale range from.75 to.91.
Mindful Attention Awareness Scale (MAAS) | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  This scale contains 15 items that describe scenes of attention deficit in daily life. Participants were required to assess the frequency of these situations based on the Likert six-point scale (1= almost always, 6= almost never). The scoring method is to directly add up the scores of all 15 items and take the average. Therefore, the score range is from 1 to 6 points. The higher the score, the higher the individual's level of attention and awareness in daily life. MAAS is a classic tool in the field of mindfulness research. It has a widely used Chinese version and has demonstrated good reliability and validity among Chinese college students. The study by Chen Siyi et al. (2012) verified the one-dimensional structure of the Chinese version of MAAS and reported its internal consistency reliability (Cronbach's α) as 0.82.
Athlete Mindfulness Questionnaire (AMQ) | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  AMQ consists of 16 items and is mainly divided into three core dimensions: Present moment attention, Awareness and Acceptance. This scale is scored using a 5-point Likert scale (for example: 1 = "Never" to 5 = "always"), with a total score range of 16 to 80 points. The higher the score, the higher the level of trait mindfulness of the athlete in the sports situation. Previous studies have shown that AMQ has good reliability and validity. In the application of sports psychology, a higher AMQ score is significantly associated with lower experience avoidance, athlete burnout and negative emotions among athletes. Meanwhile, it is positively correlated with higher well-being, flow experience and positive emotions (Zhang et al., 2015), which shows the important value of AMQ in evaluating the psychological state and potential performance of athletes.
Ryff's Scales of Psychological Well-being (18-item) | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  The scale is scored using the Likert six-point scale. Some reverse questions need to be processed first, and then the scores of the six sub-dimensions are calculated respectively, with each dimension consisting of three items. The higher the score, the higher the individual's level of psychological well-being in the corresponding dimension. The Chinese version of this scale has been widely verified. Li's (2006) research shows that the Chinese version has good reliability and validity in the sample of college students, and the internal consistency reliability (Cronbach's α) of each subscale ranges from.63 to.84
Positive and Negative Affect Scale (PANAS) | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  This study will require participants to rate the intensity of each emotional word based on their real feelings over the "past week" using a five-point Likert scale (1= very mild or none, 5= extreme). When scoring, the scores of the 10 items on each of the two subscales are added together to obtain two independent scores, each ranging from 10 to 50 points. The reliability and validity of this scale in Chinese samples are good. The study by Huang Li et al. (2003) shows that the internal consistency reliability (α) of the Chinese version of PANAS on the positive and negative subscales is 0.85 and 0.83, respectively.
Pittsburgh Sleep Quality Index (PSQI) | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  This scale contains 19 self-assessment items, which are summarized into seven core dimensions: (a) Subjective Sleep Quality; (b) Sleep Latency; (c) Sleep Duration; (d) Habitual Sleep Efficiency; (e) Sleep Disturbances; (f) Use of Sleeping Medication; And (g) Daytime Dysfunction. Each dimension is rated from 0 to 3 points. The total score is obtained by adding up the scores of all dimensions, ranging from 0 to 21 points. According to the criteria of Buysse et al. (1989), a total Score greater than 5 (Global Score > 5) is usually regarded as poor sleep quality. The reliability and validity of the Chinese version of this scale have been verified in multiple Chinese samples. For instance, Tsai et al. (2005) reported in their study in Taiwan that its internal consistency reliability (Cronbach's α) was.83, demonstrating good reliability.
Muscular Strength | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  This study adopted the 1RM test of bench press and squat. For bench presses, the testing process will strictly follow the guidelines of the National Strength and Fitness Association (NSCA) of the United States. After a thorough warm-up, participants will start with a weight close to their limit for one attempt. If the attempt is successful, give a complete rest of 3 to 5 minutes, and then increase the weight by 2.5 to 5 kilograms as appropriate for the next attempt. The entire process will involve finding the maximum weight (kg) that the individual can complete within a standard, full range of motion in 3 to 5 formal attempts. Squat to warm up and give 1 rm test process is similar to the bench press, but increase the weight of the usually after successful attempt for 5 to 10 kilograms. A successful attempt requires participants to squat until their hip joints are lower than their knee joints and stand up without assistance.
Power | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  The test data of Countermovement Jump (CMJ) and Squat Jump (SJ) will be obtained through professional Jump test pads (Just Jump System, Probotics, Inc., Huntsville, AL) It was collected in the USA. During the CMJ test, participants stand in the center of the test mat with their hands on their hips. According to the instructions, the participants quickly squatted down to an Angle of approximately 90 degrees with their knees, and then jumped up vertically with all their might without pause. For SJ, participants need to start from a static half-squat position (with the knee joint at approximately a 90-degree Angle), maintain this squat position for 2-3 seconds, and then make a vigorous vertical jump upwards. Keep both hands on your hips throughout the test. The scoring and test frequency regulations are the same as those for CMJ. The highest jump height (cm) among the three test jumps is taken as the final score.
Lane Agility Drill, LAD | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  The test was conducted in the free throw area (restricted area /Box) of the basketball court, using an electronic timing gate system (Witty SEM, Microgate, Bolzano, Italy) for precise timing. Participants start from a standing position on one side of the elbow area. Upon hearing the signal, they sprint forward to the baseline and touch the line with their feet. Then, move laterally in a defensive sliding position across the entire penalty area (4.9 meters) to the other side of the baseline and touch the line. Then, step back along the edge of the penalty area to the elbow area on that side and touch the line. Finally, move laterally across the entire free-throw line (4.9 meters) in a defensive sliding position, return to the starting point, and complete the test after the body fully passes through the timer. Each participant will take two valid tests, and the shortest time (in seconds) will be recorded as the final score.
Linear Sprints | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  To evaluate the basic running speed, a 20-meter straight-line sprint test will be adopted. An electronic timing gate system is used, with a pair of photoelectric sensors set up at the starting point and the 20-meter finish line respectively. Participants start from a position 30 centimeters behind the starting line and, upon hearing the signal, sprint forward with all their might. The system will automatically record the time (in seconds) required to complete 20 meters. Each participant will take two tests with a 3-5 minute break in between, and the best score will be taken (Stojanovic et al., 2019).
Sport-Specific Endurance | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  This study will use the Yo-Yo intermittent Recovery Test Level 1 (YYIR1). Participants will wear a Polar H10 heart rate band (Polar Electro Oy, Kempele, Finland) on their chest. The heart rate band will pair with the Polar Team app on the researchers' handheld iPad via Bluetooth for real-time data monitoring. At the beginning of the test, the participants stood at point B. According to the pre-recorded audio signal (beep), participants need to sprint to point C and run back to point B before the next signal rings. After completing each 40-meter shuttle run, participants will have A 10-second dynamic recovery time. During this period, they need to jog to point A and then return to point B to prepare for the next shuttle run. The intervals of audio signals will be systematically and gradually shortened according to the standardized YYIR1 protocol, thereby requiring participants to constantly increase their running speed to keep up with the rhythm.
Sit and Reach Test | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  The Sit and Reach Test will use the standardized measurement box (Lafayette Instrument Company, Lafayette, IN, USA). Before the test, participants will do a brief warm-up and complete two slow, informal stretching exercises. During the formal test, participants need to remove their shoes and socks, sit on the ground, keep their legs fully extended at the knee joints, and place the soles of their feet flat on the vertical surface of the measurement box. Participants need to place both hands with the palms facing down, one hand on top of the other, and the fingertips aligned. According to the instructions, participants need to slowly and smoothly lean their upper bodies forward and push their fingertips as far forward as possible along the measuring ruler. No bouncing or rapid movements are allowed during the process.Each participant will take three valid tests with a short break in between. The best score among the three measurements will be used as the final analysis data.
Single-Leg Stance Test | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  During the test, participants need to place their hands on their waists and lift the non-supporting leg so that their ankles do not touch the supporting leg. The test consists of two conditions: First, an "eye-opening" test is conducted, where participants need to focus on a fixed target point about 3 meters ahead. Then, a "closed-eye" test was conducted. Participants first opened their eyes and stood steadily. Once they were stable, they closed their eyes according to the instructions, and the timing began immediately. The test ends immediately when the supporting foot moves in any way (such as jumping or rotating), the lifted foot touches the ground, or both hands leave the hips, and the duration (in seconds) is recorded. Each leg will be tested three times under each condition (open eyes/closed eyes), with a short break between each test.
Back Scratch Test | From enrollment to the end of intervention at 8 weeks, and a 3 months follow up
  After a brief shoulder warm-up, the participants took a standing position. The researchers will guide them to raise one arm (such as the right hand) over the same shoulder, with the palm facing and touching the back, and the fingers straight and extending as downward as possible along the midline of the spine. At the same time, wrap the other arm (left hand) from under the body to behind the back, keep the back of the hand close to the back, straighten the fingers and stretch them up as much as possible, and try to make the middle fingers of both hands touch or overlap each other. Researchers will use a standard measuring ruler to precisely measure the distance between the tips of the middle fingers of both hands.Two tests will be conducted on each side, and the best score (in centimeters) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: SiMan LEI, Doctoral, Principal Investigator — University of Macau
Locations (2):
- Macau (2):
  - UM Sports Complex (N8) , Avenida da Universidade Taipa, Macau, China, Macao
  - University of Macau, Macao

IPD SHARING:
Plan to Share IPD: No